CLINICAL TRIAL: NCT04980521
Title: Promoting Radon Testing Via Smartphone App: A Clinical Trial in a High Radon State
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Dakota (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Soojung Kim, Associate Professor, University of North Dakota
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CTR radon DaCCoTA; 5U54GM128729-05 (NIH)
Record Dates: First submitted 2021-07-06; First posted 2021-07-28 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Print brochures (Placebo Comparator): Participants assigned to the print brochure group will receive three educational print brochures about radon published by EPA via postal mails for three months (one per each month).
  Interventions: Other: Print brochure
- The radon app (Experimental): Participants assigned to the radon app group will be asked to use the radon app for three months where they will be exposed to mobile friendly educational content that is created from educational print brochures about radon published by EPA.
  Interventions: Other: The radon app

INTERVENTIONS:
Other: The radon app — Participants will be asked to use the radon app.
  Arms: The radon app
Other: Print brochure — Participants will receive print brochures.
  Arms: Print brochures

SUMMARY:
This research will compare (1) the effectiveness of a mobile radon-education app (vs. traditional brochures) and (2) that of the radon app with in-app reminders (vs. the radon app without in-app reminders and the no app use with postal reminders) to increase radon awareness and testing among North Dakotans. The prevalence of exceptionally high levels of residential radon in North Dakota (ND), coupled with public's poor understanding of this hazard, is a critical public health problem.

ELIGIBILITY:
Inclusion Criteria:

* The principal eligibility criterion is that participants own a smartphone.

Exclusion Criteria:

* The principal exclusion criterion is previous testing for radon within the past two years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Soojung Kim, Principal Investigator — University of North Dakota
Locations (1):
- University of North Dakota, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim S, Chiu T, Klug MG, Schmitz D, Schwartz GG. Interventions to promote home radon testing: A randomized clinical trial of a smartphone app vs. printed brochures. Cancer Med. 2023 Jan;12(2):2027-2032. doi: 10.1002/cam4.4988. Epub 2022 Jun 28. PMID 35762397

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Some participants did not meet the eligibility criteria. They enrolled the study, but before random assignment began, they were directed to the end of the study due to not being eligible.
Period: Overall Study
Arm/Group | Print Brochures | The Radon App
Started | 68 | 70
Completed | 50 | 57
Not Completed | 18 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Print Brochures | The Radon App | Total
Number analyzed (Participants) | 68 | 70 | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16 | 24 | 40
  Between 18 and 65 years | 52 | 46 | 98
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant in the radon app group didn't provide sex/gender information. One participant in the brochure group also didn't provide sex/gender information.
  Participants
    number analyzed (Participants) | 67 | 69 | 136
    Female | 43 | 44 | 87
    Male | 24 | 25 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 57 | 58 | 115
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 68 | 70 | 138
Radon testing history [Count of Participants; unit: Participants] | 18 | 13 | 31

OUTCOME MEASURES:

1. Primary Outcome: Ordering a Free Radon Test Kit
Description: The rate at which participants order a free radon test kit
Time Frame: Through the study completion - 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Print Brochures | The Radon App
Number analyzed (Participants) | 68 | 70
Participants | 9 | 29

2. Primary Outcome: Using the Radon Test Kit
Description: The rate at which participants use the radon test kit to test their houses
Time Frame: Through the study completion - 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Print Brochures | The Radon App
Number analyzed (Participants) | 9 | 29
Participants | 2 | 2

3. Secondary Outcome: Change From Baseline Radon Knowledge at 3 Months
Description: Radon knowledge was measured by the number of accurate responses to 20 True-False statements in T1 (baseline) and T2 (at 3 months), as used in Kim, Brewster, and Schwartz (2020) (PMID: 32321499). The response options were: "true," "false," and "I don't know." Participants' responses to each statement were then re-coded to 1 ("correct") or 0 ("incorrect" or "I don't know"). After that, two radon knowledge index variables (continuous) were created by summing participants' responses to each statement in T1 (baseline) and T2 (at 3 months). Thus, two radon knowledge scores can range from 0-20 with higher scores indicating better knowledge.
Time Frame: Change from baseline knowledge level to the completion of study at 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Print Brochures | The Radon App
Number analyzed (Participants) | 50 | 57
units on a scale | -0.4 (1.3) | 2.2 (1.2)

ADVERSE EVENTS:
Time Frame: 6 months.
Arm/Group | Print Brochures | The Radon App
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/70
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/70
Other Adverse Events (participants affected / at risk) | 0/68 | 0/70

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT04980521/Prot_SAP_000.pdf
  • Informed Consent Form (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT04980521/ICF_001.pdf